CLINICAL TRIAL: NCT00214474
Title: Improving Diabetes Efforts Across Language and Literacy (IDEALL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Collaborators: The Commonwealth Fund (Other); California HealthCare Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R21HS014864-01 (AHRQ)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes
Keywords: Disease Management; Health Literacy; Telephone Care; Group Medical Visits; Type 2 Diabetes; Access to Care; Technology; Language Barriers
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ATSM Intervention (Active Comparator): ATSM Intervention: Automated Telephone Self-Management Support
  Interventions: Behavioral: ATSM Intervention
- GMV Intervention (Active Comparator): GMV Intervention: Group Medical Visits
  Interventions: Behavioral: GMV Intervention
- Usual Care (No Intervention): Usual Care: Standard care for diabetic patients

INTERVENTIONS:
Behavioral: ATSM Intervention — Participants randomized to ATSM Intervention received weekly, automated (pre-recorded) telephone calls over 39 weeks (9 months). Patient responses triggered either immediate, automated health education messages and/or subsequent nurse phone follow-up.
  Other Names: ATSM: Automated Telephone Self-Management Support
  Arms: ATSM Intervention
Behavioral: GMV Intervention — GMV Intervention involved 90-minute monthly sessions over 9 months, involving 6-10 participants, co-facilitated by a primary care physician and health educator.
  Other Names: GMV: Group Medical Visits
  Arms: GMV Intervention

SUMMARY:
The IDEALL Project (Improving Diabetes Efforts Across Language and Literacy) is a 3-arm randomized controlled trial to explore contextual factors at the patient, clinician, and organizational level of two patient self-management support strategies. A communication technology-based intervention (automated telephone diabetes management) and an interpersonally-oriented intervention (group medical visits)will be compared to usual care for their ability to improve diabetes outcomes among vulnerable populations in 4 safety-net health centers in the University of California, San Francisco (UCSF) Collaborative Research Network.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* have type 2 diabetes
* have a HbA1c equal to or > 8.0%
* must speak English, Spanish, or Cantonese.

Exclusion Criteria:

* Dementia
* Psychosis/Schizophrenia
* End Stage Renal Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2002-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Changes in Diabetes Self-management Behaviors as Measured by Summary of Diabetes Self-Care Activities (SDSCA) Scale | Baseline and 1 year
  The Summary of Diabetes Self-Care Activities (SDSCA) Measure is a brief self-report questionnaire on diabetes self-management behaviors. The questionnaire assesses the frequency with which a patient followed a diabetes routine over the prior 7 days in five domains: diet, exercise, blood-glucose testing, foot care, and medication adherence. Based on SDSCA measure's author's recommendations, two separate scores can be derived: a Diabetes Self-management Behaviors score and a Self-reported Medication Adherence score. The Diabetes Self-management Behaviors score is used in this study. For this score, all items pertaining to diet, exercise, blood glucose testing, and foot care are averaged. The result is an average score between 0 and 7 with higher score indicating better diabetes self-management behavior. Change is calculated as 1-year score minus baseline score.
Changes in Minutes of Moderate Physical Activity | Baseline and 1 year
  A measure of patients' physical activity is ascertained by asking patients the following question: "In the last 7 days, how many total minutes or hours did you do physical activity? Like walking, house cleaning or gardening." Number of minutes may range from 0 to 10080, with greater number of minutes indicating more physical activity.
Changes in Minutes of Vigorous Exercise | Baseline and 1 year
  A measure of patients' vigorous exercise is ascertained by asking patients the following question: "In the last 7 days, how many total minutes or hours did you do the kind of exercise that makes you breathe hard, such as swimming, walking fast, or biking?" Number of minutes may range from 0 to 10080, with greater number of minutes indicating more vigorous exercise.

SECONDARY OUTCOMES:
Changes in Patient Assessment of Chronic Illness Care (PACIC) | Baseline and 1 year
  The Patient Assessment of Chronic Illness Care (PACIC) is a 20-item patient report instrument that measures patients' perspectives on the structure of their care and collects patient reports on the extent to which they have received specific clinical services and actions during the past year that are aligned with the Chronic Care Model. The scale is intended to assess the receipt of care that is patient-centered, proactive, planned and includes collaborative goal setting, problem-solving and follow-up support. Each instrument item is scored on a 5-point scale ranging from 1 to 5 with higher score indicating better care. Scores are transformed to a 100-point scale and averaged across all items to create a total scale score. Change is calculated as 1-year score minus baseline score.
Changes in Diabetes Self-efficacy as Measured by Diabetes Quality Improvement Project's Patient Self-Management Scale | Baseline and 1 year
  The Patient Self-Management Scale was derived from a questionnaire used in the Diabetes Quality Improvement Project. The scale is designed to reflect patients' assessment of their ability to manage aspects of diabetes self-care in 5 separate areas (medication, diet, exercise, blood glucose monitoring, and foot care). Respondents are asked how difficult over the past year has it been to follow exactly as their doctor who takes care of their diabetes suggested. Possible scores for each scale item range from 0 to 100 with higher score indicating more self-efficacy. Total scale score is calculated as the average across all items. Change is calculated as 1-year score minus baseline score.
Changes in Interpersonal Processes of Care (IPC) Scale | Baseline and 1 year
  The Interpersonal Processes of Care (IPC) captures patient reports of providers' communication over the prior year. The scale is intended to measure patients' assessment of providers' communication within 3 broad domains: communication (e.g., lack of clarity), decision making (e.g., patient-centered decision making), and interpersonal style (e.g., friendliness). Each instrument item is scored on a 5-point scale ranging from 1 to 5. Scores are transformed to a 100-point scale and averaged across all items to create a total scale score. Higher total scores indicate better communication. Change is calculated as 1-year score minus baseline score.
Changes in the Physical Component Summary of the SF-12 Health Survey | Baseline and 1 year
  The SF-12 Health Survey (SF-12) is a 12-item short-form survey used to measure health status and monitor health outcomes. The survey asks about various health aspects, including physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health (psychological distress and psychological well-being). Two summary measures are derived: the Physical and the Mental Health Component Summary. For each component summary, survey items were weighted and summed to create a summary score between 0 and 100 with higher score indicating better functioning and outcome. Change is calculated as 1-year score minus baseline score.
Changes in the Mental Component Summary of the SF-12 Health Survey | Baseline and 1 year
  The SF-12 Health Survey (SF-12) is a 12-item short-form survey used to measure health status and monitor health outcomes. The survey asks about various health aspects, including physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health (psychological distress and psychological well-being). Two summary measures are derived: the Physical and the Mental Health Component Summary. For each component summary, survey items were weighted and summed to create a summary score between 0 and 100 with higher score indicating better functioning and outcome. Change is calculated as 1-year score minus baseline score.
Number of Days Spent in Bed Due to Health Problems | 1 year
  A measure of patients' functional status is ascertained by asking patients the following question: "In the last 30 days, how many days did your health keep you in bed all or most of the day?" Number of days may range from 0 to 30, with lower number of days indicating better functional status.
Proportion of Patients Reporting Diabetes Interference of Normal Daily Activities | 1 year
  A measure of diabetes interference on patients is ascertained by asking patients the following question: "In the last 12 months, how often has your diabetes kept you from doing your normal daily activities, such as going to work, grocery shopping, and taking care of yourself and others?" Responses consist of 6 possible options: "Always", "Almost Always", "Often", "Sometimes", "Almost Never", and "Never". These responses are grouped into 2 categories, with one category consisting of "Always", "Almost Always", and "Often" responses while the other category consists of the remaining responses. The proportion of patients reporting diabetes interference is the number of patients in the first category divided by the number of patients in the 2 categories combined.
Changes in Hemoglobin A1c Levels | Baseline and 1 year
  Hemoglobin A1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. As the average amount of plasma glucose increases, the fraction of hemoglobin A1c increases in a predictable way. This serves as a marker for average blood glucose levels over the previous months prior to the measurement. Higher amounts of hemoglobin A1c indicate poorer control of blood glucose levels and have been associated with cardiovascular disease. Change is calculated as 1-year level minus baseline level.
Changes in Systolic Blood Pressure (SBP) | Baseline and 1 year
  Systolic blood pressure is the pressure exerted on arteries and vessels by the heart when it contracts and pushes blood through the arteries to the rest of the body. Change is calculated as 1-year pressure minus baseline pressure.
Changes in Diastolic Blood Pressure (DBP) | Baseline and 1 year
  Diastolic blood pressure is the pressure exerted on the walls of the arteries and vessels in between heart beats, when the heart is relaxed and dilated, filling with blood. Change is calculated as 1-year pressure minus baseline pressure.
Changes in Body Mass Index (BMI) | Baseline and 1 year
  Body Mass Index (BMI) is a number calculated from a person's weight and height. BMI is defined as the individual's body mass divided by the square of their height. The formulae used produce a unit of measure of kg/m2. BMI provides an indicator of body fatness.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Schillinger, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Ucsf Dept of Medicine Box 1364, San Francisco, California, United States

REFERENCES:
- [Derived] Schillinger D, Handley M, Wang F, Hammer H. Effects of self-management support on structure, process, and outcomes among vulnerable patients with diabetes: a three-arm practical clinical trial. Diabetes Care. 2009 Apr;32(4):559-66. doi: 10.2337/dc08-0787. Epub 2009 Jan 8. PMID 19131469